CLINICAL TRIAL: NCT06153368
Title: Cadonilimab Plus mFOLFIRINOX as Conversion Therapy in Patients With Locally Advanced Pancreatic Cancer：A Prospective, Single-arm, Phase II Trial
Brief Title: Cadonilimab Plus mFOLFIRINOX as Conversion Therapy in LAPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kuirong Jiang, chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-566
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (Experimental): Drug：Cadonilimab 6 mg/kg，IVD，D1，Q2W Drug：mFOLFIRINOX mFOLFIRINOX（Oxaliplatin 85 mg/m2 IV over 4 hours ; Irinotecan 150 mg/m2 IV over 90 minutes ; Leucovorin(l-LV) 400 mg/m2 IV over 2 hours 5-fluorouracil 2.4 g/m2 for 46 hours continuous infusion.） on days 2 of a 14-day cycle.
  Interventions: Drug: Cadonilimab+mFOLFIRINOX

INTERVENTIONS:
Drug: Cadonilimab+mFOLFIRINOX — Cadonilimab 6 mg/kg，IVD，D1，Q2W
  +mFOLFIRINOX（Oxaliplatin 85 mg/m2 IV over 4 hours ; Irinotecan 150 mg/m2 IV over 90 minutes ; Leucovorin(l-LV) 400 mg/m2 IV over 2 hours 5-fluorouracil 2.4 g/m2 for 46 hours continuous infusion.） on days 2 of a 14-day cycle.
  Other Names: Cadonilimab+Oxaliplatin+ Irinotecan+ Leucovorin+ 5-fluorouracil

SUMMARY:
This is a prospective, single arm, single center, phase II study of cadonilimab plus mFOLFIRINOX as conversion therapy in patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Eligible patients with histologically/cytologically confirmed unresectable locally advanced pancreatic cancer (LAPC) will receive cadonilimab (6mg/kg，IVD，D1，Q2W) plus mFOLFIRINOX (oxaliplatin 85mg/m2 , D2 + leucovorin 400mg/m2 , D2 + irinotecan 150mg/m2 , D2 + 5-fluorouracil 2,400mg/m2 46h continuous infusion ) for 4 cycles (8 weeks).

After completing every 4 treatment cycles, the subjects will undergo imaging examinations of tumor lesions. If the subjects do not experience disease progression, they will continue to receive treatment until surgical resection, disease progression (RECIST 1.1), or intolerable toxic reactions occur, new anticancer drug treatment begins, withdrawal from the study, death, or loss of follow-up. All subjects who have received treatment are required to undergo efficacy evaluation every 8 weeks (± 7 days) after the start of treatment, until disease progression or study termination. After the 12th cycle of treatment, the maintenance treatment plan is to use capecitabine or S-1 combined with cadonilimab for maintenance treatment. During maintenance treatment, imaging efficacy evaluation is conducted every 12 weeks (± 7 days), and surgical resectability is still evaluated until surgical resection, disease progression (RECIST 1.1) or intolerable toxic reactions occur, new anticancer drug treatment begins, withdrawal from the study, death, or loss of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas.
2. Patients must have locally advanced pancreatic cancer (LAPC).
3. Patients must have LAPC evaluated by radiologist and/or surgeon according to either abdominal CT or MRI, or intra-operative findings.

   Locally advanced unresectable disease was defined by CT or MRI images as low-density tumor (primary and/or lymphadenopathy) with
   1. extension to the celiac axis or superior mesenteric artery,
   2. occlusion of the superior mesenteric-portal venous confluence
   3. aortic, inferior vena cava (IVC) invasion or encasement
   4. invasion of superior mesenteric vein below transverse mesocolon or unresectable after surgical exploration.

   Those who had superior mesenteric vein impingement, superior mesenteric artery abutment were defined as borderline resectable.

   Those who had superior mesenteric vein occlusion, superior mesenteric artery encasement were defined as unresectable.
4. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 8.2 for the evaluation of measurable disease.
5. Age ≥18years and ≤75 years.
6. Eastern Cooperative Oncology Group performance score of 0 or 1; see Appendix A.
7. Patients must have normal organ and marrow function
8. Patients who present with jaundice will be allowed to enroll after control with temporary or permanent internal/external drainage.
9. The effects of study agents on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with distant metastases are not eligible.
2. Patients with endocrine or acinar pancreatic carcinoma.
3. Patients may be receiving any steroid, immunologic or other investigational agents within 4 weeks prior to enrollment.
4. Patients who have had prior chemotherapy or radiotherapy are not eligible.
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents used in the study.
6. Patients who have above grade II peripheral neuropathy.
7. Patients who had non-curable second primary malignancy within five years, except for non-melanoma skin cancer.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant women are excluded from this study because the study agents has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
10. Those who are immuno-compromised or receiving immuno-suppressive therapy are excluded from the study because of increased risk of lethal infections and possible pharmacokinetic interactions with study agent administered during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-19 (Estimated); Primary Completion 2024-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  ORR is defined as the percentage of participants who have a confirmed complete response or partial response according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to two years
  PFS is defined as the time from enrollment of the trial to the first documented disease progression or death due to any cause.
Overall survival (OS) | Up to two years
  The duration from the date of recruitment to the date of death from any cause.
Adverse events (safety) | Up to two years
  Adverse events (safety ) will be evaluated according to the NCI CTCAE Version 5.0.The number and severity of treatment-related side effects, including AE and SAE, will be recorded during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rong K Jiang, MD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.